CLINICAL TRIAL: NCT03089190
Title: SLIM8 - Acute Effects of DC7-2 on Appetite
Brief Title: Acute Effects of DC7-2, a Meat Derived Octapeptide, on Appetite
Acronym: SLIM8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arne Astrup (Other)
Responsible Party: Sponsor-Investigator, Arne Astrup, Head of Department, Professor MD DMSc, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B330
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Appetite; Lack or Loss, Nonorganic Origin
Keywords: Appetite; Satiety; Energy intake; Hunger; Peptide; Encapsulation

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized crossover design with four arms including three experimental conditions and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DC7-2 alone (Active Comparator): Administration of DC7-2, a meat-derived octapeptide.
  Interventions: Dietary Supplement: DC7-2
- DC7-2 + potato protein isolate (Active Comparator): Administration of DC7-2, a meat-derived octapeptide, combined with potato protein isolate that protects DC7-2 from degradation in the GI tract.
  Interventions: Dietary Supplement: DC7-2 + potato protein isolate
- Potato protein isolate + placebo (Active Comparator): Administration of potato protein isolate combined with inactive whey protein as placebo.
  Interventions: Dietary Supplement: Potato protein isolate
- Placebo (Placebo Comparator): administration of inactive whey protein
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: DC7-2 — Effects on appetite
  Arms: DC7-2 alone
Dietary Supplement: DC7-2 + potato protein isolate — Effects on appetite
  Arms: DC7-2 + potato protein isolate
Dietary Supplement: Potato protein isolate — Effects on appetite
  Arms: Potato protein isolate + placebo
Dietary Supplement: Placebo — Inactive whey protein, not expected to affect appetite.
  Arms: Placebo

SUMMARY:
A double-blind, randomized crossover design with four arms including three experimental conditions and placebo will be applied. After having successfully completed screening procedures, eligible participants will be invited to four separate test days. The test days are separated with at least 7 days, however 4 days can be accepted for logistical reasons. During the entire course of the study, participants must remain weight stable and not change their diet or physical activity level. Significant changes in diet, physical activity level (evaluated by the sub-investigator) or weight change ±3 kg over the course of the study (from screening to completion of the last test day) results in exclusion of that subject.

DETAILED DESCRIPTION:
For standardization, participants will be asked avoid excessive alcohol consumption (not above 1 unit and no alcohol at all from 8 pm the night before the test days) and intense physical activity 48 hours prior to the test day. Also, they will be asked to consume a standardized meal at home no later than 8 pm the night before the test days. This meal is prepared and delivered by the department.

Furthermore, the participants must arrive at the study facilities in the morning after an overnight fast (from 10 pm) using non strenuous means of transportation.

Over the course of the study (from screening (visit 1) to completion of the last test day (visit 5)), participants are not allowed to change body weight (±3 kg), diet or physical activity level (as judged by the sub-investigator). The participants will be weighed and asked about compliance with additional standardization before initiating each test day. Possible in-compliance with the standardization will be judged by the sub-investigator whether to result in rescheduling of the visit or to be recorded as a protocol deviation.

Participants arrive at the study facility in the morning. Compliance with standardization is controlled along with registration of possible adverse events and use of concomitant medications. During the test days, participants are settled together with other participants, but separated at individual tables. During the meals, participants are settled into individual feeding cubicles, where they cannot see each other and are instructed not to talk to each other. Visual analogue scales (VAS') will be completed for measurement of fasting subjective appetite levels.

The test products (capsules) will be provided prior to a standardized fixed breakfast, prior to a standardized fixed mid-morning snack and prior to an ad libitum meal. Immediately before and after each episode of capsules and food consumption and at 30 minutes intervals, VAS' will be completed. Energy intake will be calculated from the ad libitum meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Age between 18 and 65 years
* BMI between 27-35 kg/m2

Exclusion Criteria:

* Vegetarians
* Participants unable to consume or known to get nausea from consuming capsules
* Participants not able to comply with the study protocol, including consumption of the specific study foods (pictures of study foods shown at screening)
* Any known food allergies or food intolerance likely to affect the present study
* Weight change of ±3 kg two months prior to the study
* Vigorous physical activity more than 5 hours/week
* Alcohol intake above the recommendations from the Danish Health and Medicines Authority (>14 units/week)
* Substance abuse
* Smoking, smoking cessation within the past 3 months or nicotine use (electronic cigarettes, gum etc.). Irregular smokers accepted
* Use currently or within the previous 3 months of any medication or supplements known to affect appetite or body weight as judged by the investigators
* Chronic diseases (e.g. cancer, thyroid disease, heart disease, diabetes, neurological disorders, or sleep disorders) or other relevant health problems as judged by the investigators
* Simultaneous or within the past month participation in other clinical studies
* Participant's general condition contraindicates participating in the study, as judged by the investigators or the medical expert

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Selfreporting
Enrollment: 32 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Energy intake | 360 min
  Assessment of ad libitum energy intake when exposed to one of the test products

SECONDARY OUTCOMES:
Subjective appetite sensations | Six hours during each test day between test day 1, 2, 3, and 4 (acute effect)
  Evaluations of each of the subjective appetite sensations assessed by visual analogue scale (VAS) (satiety, fullness, hunger, prospective food consumption, thirst)

OTHER OUTCOMES:
Palatability of meals | Directly after consumption of the three meals at all four test days
  All three meals are rated for their palatability e.g. smell, taste and appearance
Subjective assessments of nausea and general wellbeing | Six hours during each test day between test day 1, 2, 3, and 4 (acute effect)
  VAS assessments for nausea and general wellbeing throughout the study test day

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, MD DMSc, Principal Investigator — Department of Nutrition, Exercise and Sports, Research Centre Opus, University of Copenhagen, Rolighedsvej 26, 1958 Frederiksberg C
Locations (1):
- Department Of Human Nutrition, Faculty of Science, University of Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared